CLINICAL TRIAL: NCT06290739
Title: Development and Validation of a Machine-learning Model to Predict Lymph Node Metastasis of Intrahepatic Cholangiocarcinoma: a Retrospective Cohort Study.
Brief Title: A Machine-learning Model to Predict Lymph Node Metastasis of Intrahepatic Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiwei Huang, Dr., Sichuan University
Other Study IDs: JHuang886
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Intrahepatic Cholangiocarcinoma; Machine Learning
Keywords: Intrahepatic Cholangiocarcinoma; machine learning; prognosis; online calculator
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intrahepatic cholangiocarcinoma patients who underwent lymph nodes dissection
  Interventions: Procedure: lymph nodes dissection
- Intrahepatic cholangiocarcinoma patients who didn't undergo lymph nodes dissection

INTERVENTIONS:
Procedure: lymph nodes dissection — Whether lymph nodes dissection should be performed on curative-intent hepatectomy for intrahepatic cholangiocarcinoma is still debated.
  Groups: Intrahepatic cholangiocarcinoma patients who underwent lymph nodes dissection

SUMMARY:
The object of this study is to develop a model for prediction of lymph node metastasis among intrahepatic cholangiocarcinoma (ICC) patients. Intrahepatic cholangiocarcinoma is the second most common kind of primary liver cancer, accounting for approximately 10%-15%. There is a lack of agreement regarding the necessity of performing lymph node dissection (LND) in patients with ICC. Currently, the percentage of LND is below 50%, and the rate of sufficient LND (≥6) has plummeted to less than 20%. Consequently, a large proportion of patients are unable to acquire LN status, which hinders the following systematic treatment strategies after surgery:. Therefore, our objective is to construct a LN metastasis model utilizing machine learning techniques, including patients' clinical data and pathology information, with the goal of offering a reference for patients who have not undergone LND or have had inadequate LND.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients who were confirmed with intrahepatic cholangiocarcinoma 2. curative-intent hepatectomy 3. Without concurrent extrahepatic disease

Exclusion Criteria:

* 1.Patients lacking complete pathology information, 2. Patients who didn't get curative resection 3.Patients with concurrent extrahepatic disease or had missing follow-up data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The data was collected from patients who underwent curative-intent hepatectomy and were diagnosed with ICC pathologically. The data was collected from the hepato-biliary and pancreatic department of West China Hospital, SCU, between the periods of January 2010 to December 2016 and January 2019 to October 2023.
Sampling Method: Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2010.01-2019.01
  Overall survival (OS) refers to the duration between the commencement of surgery and the patient's demise due to any reason.

SECONDARY OUTCOMES:
Disease free survival | 2010.01-2019.01
  Disease-free survival (DFS) refers to the period of time from the date of surgery until the occurrence of a relapse either within or outside the liver.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Liver Surgery and Liver Transplantation Center, West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
The data that supports the findings of this study is available from the corresponding author upon reasonable request.